CLINICAL TRIAL: NCT02148978
Title: DPP-IV Inhibition in Patients With Cystic Fibrosis
Brief Title: Cystic Fibrosis Related Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ram Weiss (Other)
Responsible Party: Sponsor-Investigator, Ram Weiss, Professor, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0016-14-HMO
Record Dates: First submitted 2014-05-15; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — saxagliptin

ARMS (1):
- Saxagliptin administration (Experimental): Saxagliptin Administration- The participants in this study will undergo an OGTT (Oral Glucose Tolerance Test) at recruitment and then will start treatment with the DPP IV inhibitor- Saxagliptin. After 6 weeks of treatment the participants will return to perform a second OGTT.
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin — The participants in this study will undergo an OGTT at recruitment and then will start treatment with the DPP IV inhibitor- Saxagliptin at a dose between 2.5- 5mg a day. After 6 weeks of treatment the participants will return to perform a second OGTT.

SUMMARY:
Cystic Fibrosis (CF) is a chronic disease characterized by recurrent pulmonary infections and exocrine pancreatic insufficiency. The vast majority of patients with CF will develop pancreatic endocrine insufficiency over time manifested as altered glucose metabolism. The presence of overt diabetes in patients with CF is associated with adverse clinical outcomes.

The underlying pathophysiology of cystic fibrosis related diabetes (CFRD) is still a matter of investigation. In addition to localized tissue damage developing similar to that of the exocrine pancreas, additional mechanisms may be involved. The investigators have recently shown that insulin secretion in patients with CF is significantly altered prior to the development of diabetes. This phenomenon is associated with reduced secretion of gut derived incretins (specifically GIP). The blunting of incretin induced insulin secretion (whether due to a deranged interaction of gastrointestinal contents with enterocytes resulting in reduced secretion or due to rapid clearance of such peptides) may be a major underlying driver of altered glucose metabolism in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* No diabetes based on screening OGTT
* No C/I for use of the medications
* Normal kidney function
* Willing and able to participate

Exclusion Criteria:

* Use of anti-hyperglycemic medications
* Acute illness or infection at enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
glucose tolerance after treatment with Saxagliptin | The outcome will be measured at 2 timepoints. at baseline and 6 weeks after Saxagliptin treatment
  Bloods taken during the OGTT will be analyzed for Glucose, Insulin, C-peptide and glucagon levels. Gut hormone levels and incretins will also be valued.

CONTACTS AND LOCATIONS:
Overall Officials: Limor Marko, MSc, Principal Investigator — Hebrew University; Eitan Kerem, MD, Principal Investigator — Hadassah Har Hazofim; Karen Hershkop, PhD, Principal Investigator — Hebrew University
Locations (1):
- Hadassah Har Hazofim, Jerusalem, Israel